CLINICAL TRIAL: NCT06413862
Title: Efficacy and Safety of Ciprofol Versus Propofol in Patients Undergoing Painless Hysteroscopy
Brief Title: Ciprofol Versus Propofol in Patients Undergoing Painless Hysteroscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baoding First Central Hospital (Other)
Responsible Party: Principal Investigator, Lei Zhu, Chief Physician, Baoding First Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ciprofol in hysteroscopy
Record Dates: First submitted 2024-05-07; First posted 2024-05-14 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Painless Hysteroscopy
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol group (ciprofol combined with alfentanil) (Experimental)
  Interventions: Drug: Ciprofol
- Propofol group (propofol combined with alfentanil) (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ciprofol — The experimental group was slowly injected with ciprofol for 30 seconds (0.4mg/kg, Haisike Pharmaceutical Co., Ltd., Liaoning, China, batch number 20220911).
  Arms: Ciprofol group (ciprofol combined with alfentanil)
Drug: Propofol — The control group was slowly injected with propofol for 30 seconds (2mg/kg, Guorui Pharmaceutical Co., Ltd., Sichuan, China, batch number 22102914).
  Arms: Propofol group (propofol combined with alfentanil)

SUMMARY:
Ciprofol exhibits comparable efficacy to that of propofol, and is associated with less injection pain rate, fewer adverse events, higher patient satisfaction, and more stable hemodynamics when used for general anesthesia during the painless hysteroscopy.

DETAILED DESCRIPTION:
In this study, we found that sedation success rate was 100% in both ciprofol group and propofol group during the painless hysteroscopy. The incidence rate of injection pain and the intensity of pain in the ciprofol group were significantly lower than the propofol group. Also, the ciprofol group had lower incidence rate and severity level of adverse events and higher patient satisfaction. In addition, SBP, DBP, and MAP values in propofol group were found to be significantly lower than those in ciprofol group at the time of cervical dilation and of consciousness recovery.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years old;
2. undergoing hysteroscopy examination and requiring intravenous anesthesia;
3. American Society of Anesthesiologists (ASA) physical status I to II;
4. without communication difficulties, and able to cooperate with intervention implementation;
5. participating in this trial voluntarily, and signing an informed consent form;

Exclusion Criteria:

1. with contraindications for hysteroscopy examination (such as cervical stenosis, difficulty in cervical dilation, reproductive tract infections such as vaginitis and cervicitis) or allergies to the intended anesthetic drugs;
2. with severe cardiac insufficiency, liver and kidney dysfunction, and other major diseases;
3. with a history of uterine surgery within the past three months;
4. body temperature above 37.5 ℃ before the anesthesia;
5. long-term use of sedative or analgesic drugs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2024-09-09 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Injection pain | 24 hours within hysteroscopy
  The injection pain was defined as the pain reported verbally by patients during the first injection of the investigational drugs (ciprofol or propofol). The Numerical Rating Scale (NRS) was used to evaluate the pain level. The anesthesiologist asks the patient during the first injection of the investigational drug (ciprofol or propofol), "Do you feel arm pain from the injection? Patients who answered "yes" was asked to describe the level of the pain (a score of 0 to 10 indicated "painless" to "unbearable pain"). The pain level was divided into painless (0 points), mild pain (1-3 points), and moderate to severe pain (4-10 points).

SECONDARY OUTCOMES:
Sedation success rate | 24 hours within hysteroscopy
  No more than 5 supplementary doses within 15 minutes
Anesthesia success rate | 24 hours within hysteroscopy
  the absence of any alternative sedatives/anesthetic drugs after the initial administration of the investigational drugs
time for successful anesthesia induction | 24 hours within hysteroscopy
  the time from starting the administration of investigational drugs to the MOAA/S score ≤ 1
recovery time | 24 hours within hysteroscopy
  the time from the last administration of investigational drugs to awaken
use of rescue drugs | 24 hours within hysteroscopy
  ephedrine, atropine
times of supplementing ciprofol or propofol | 24 hours within hysteroscopy
  times of supplementing ciprofol or propofol
adverse events | 24 hours within hysteroscopy
  nausea, vomiting, hypoxemia (blood oxygen saturation < 90% and lasting > 30 seconds), bradycardia (heart rate < 55 beats/minute), hypotension (systolic blood pressure reduced by 20% compared to baseline), body movement (patient's unconscious limb movements) during the examination
severity level of adverse events | 24 hours within hysteroscopy
  graded based the National Cancer Institute Common Terminology Criteria for the Classification of Adverse Events (CTCAE) version 5.0, and divided into grade 1 (mild), grade 2 (moderate), grade 3 (severe or medically significant but not immediately life threatening), grade 4 (events with life-threatening consequences needing urgent intervention), grade 5 (death related to the adverse events)
patient satisfaction | 24 hours within hysteroscopy
  using a 10-point scale, with 1 point indicating extreme dissatisfaction and 10 points indicating very satisfied
comparison of vital signs before and after administration | 24 hours within hysteroscopy
  The systolic blood pressure in mmHg, diastolic blood pressure in mmHg, mean arterial pressure in mmHg, blood oxygen saturation in %, and heart rate in bpm were recorded before anesthesia induction (T0), after anesthesia induction (T1), at cervical dilation (T2), and at consciousness recovery (T3)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhu, Principal Investigator — the First Central Hospital of Baoding

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li A, Li N, Zhu L, Xu Z, Wang Y, Li J, Zhang G. The efficacy and safety of ciprofol versus propofol in patients undergoing painless hysteroscopy: a randomized, double-blind, controlled trial. BMC Anesthesiol. 2024 Nov 12;24(1):411. doi: 10.1186/s12871-024-02787-0. PMID 39533194